CLINICAL TRIAL: NCT02798497
Title: Panton Valentine Leucocidin : Independent Severity Factor of Staphylococcus Aureus Pneumonias
Brief Title: Panton Valentine Leucocidin
Acronym: PVL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010.625
Record Dates: First submitted 2016-05-27; First posted 2016-06-14 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Staphylococcus Aureus Pneumonias
Keywords: PVL; Pneumonias; Staphylococcus aureus
MeSH Terms: conditions — Pneumonia, Staphylococcal; Pneumonia; Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- staphylococcus aureus PVL- (Other): patients with staphylococcus aureus PVL-
  Interventions: Other: Serum and Blood samples
- staphylococcus aureus PVL+ (Other): patients with staphylococcus aureus PVL+
  Interventions: Other: Serum and Blood samples

INTERVENTIONS:
Other: Serum and Blood samples

SUMMARY:
Staphylococcus aureus expresses a variety of virulence factors, including Panton Valentine leukocidin (PVL), a cytotoxin. PVL is specifically associated with primary skin and soft-tissue infections and severe necrotizing pneumonia (Gillet et al. Lancet, 2002;359:753-9). PVL-positive S. aureus pneumonia is often preceded by influenza-like symptoms, and is mainly characterized by hemoptysis, pleural effusion, rapid onset of acute respiratory distress, leukopenia and a high fatality rate (65%) (Gillet et al. Lancet, 2002;359:753-9). Ten year after the first description of this disease and a number of controversies in the scientific literature, the question arise as to whether PVL remains an independent factor of severity in S.aureus pneumonia. In addition, numerous questions remain unanswered yet; these are:

* (i) which factors, including treatment regimen, are associated with favourable outcome?,
* (ii) what is the susceptibility toward antibiotics of strains associated with this disease ?
* (iii) is there any genetic susceptibility of the host to explain both the rarity, and the explosive presentation of the disease ? To address the above questions a prospective observational study at the nationwide level will be set up. All French hospitals will be invited to describe the clinical features of all new cases of S. aureus community-acquired pneumonia with severity criteria, regardless PVL production. The study will include an investigation of a possible innate immune dysfunction in collaboration with the INSERM-U550 (Génétique Humaine des Maladies Infectieuses, Faculté Necker, Paris). Hence, in addition to collecting clinical and biological data from all pneumonia cases as well as all strains of S. aureus isolated, the patients with PVL-positive pneumonia will be sampled for immune genetic studies (ORFeome sequencing and functional studied)

ELIGIBILITY:
Inclusion Criteria:

* 2-month-old patient at minimum and weighing at least 5 kg
* Informed consent
* Subjects affiliated (or beneficiary) to a national medical insurance
* Presence of clinical, biological and radiological signs of pneumopathy to S. aureus whose clinical state justifies a hospitalization in a ICU or in a reanimation
* Presence of PVL- positive S.aureus producer (for immunogenetic study)

Exclusion Criteria:

* Patients infected by the HIV
* Patients hospitalized for more than 48 hours at the time of the diagnosis of pneumonia,
* Patients hospitalized during the previous three months excepted outpatients

Ages: 2 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
The survival of the patients according to the character PVL+ or PVL- of the isolated Staphylococcus aureus strains | After hospitalisation, an average of 21 days
  Percentage of alive patients after the length of stay in hospitalisation

SECONDARY OUTCOMES:
Gravity Scores : Composite measure between the IGS2 and SOFA scores for an adult and between PIM2 and PLEOD scores for a child | At admission at Reanimation Unit or ICU, at 24 h after admission and 7 days after admission
length of stay in Reanimation and ICU | number of days in Reanimation and ICU
  After hospitalisation, an average of 21 days
length of stay in hospitalization | After hospitalisation, an average of 21 days
Number of participants with presence of a genetic predisposition of Mendelian type or polymorphic character among the patients presenting a PVL+ necrotizing pneumonia (for immunogenetic study) | at maximum 6 days after Sampling of blood and of serum
  genomic analysis an immunologic tests

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Références des Staphylocoques Centre de Biologie et Pathologie Est 59 bd Pinel, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] As designed, the study enrolled a cohort of 154 evaluable patients. In the adult subgroup, there was a balanced distribution between pneumonia caused by Staphylococcus aureus that was Panton-Valentine leukocidin (PVL)-positive and PVL-negative. This balanced allocation will enable a refined assessment of the PVL effect in this condition. Preliminary results appear to support the working hypothesis (mortality 45% in PVL-positive vs 26.3% in PVL-negative cases; p < 0.05). In addition, biospecimens were collected from 98 patients for subsequent genetic analyses.